CLINICAL TRIAL: NCT06097845
Title: Transcranial Ultrasound Via Sonolucent Cranioplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Netanel Ben-Shalom, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-0873
Record Dates: First submitted 2023-09-19; First posted 2023-10-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cranioplasty; Sonolucent Cranioplasty; Reconstructive Cranioplasty
Keywords: Transcranial Ultrasound; SOC ultrasound; PMMA implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcranial Ultrasound (Experimental): Ultrasound imaging will be performed by clinicians using FDA-approved ultrasound devices currently used in routine clinical practice.
  Interventions: Diagnostic Test: Transcranial Ultrasound

INTERVENTIONS:
Diagnostic Test: Transcranial Ultrasound — Patients who underwent reconstructive sonolucent cranioplasty will receive standard of care postoperative imaging (i.e. CT, MRI) in addition to ultrasound imaging. Ultrasound imaging will be performed by clinicians using FDA-approved ultrasound devices (GE Venue Go, Fujifilm Sonosite X-Porte, GE Volusion E10 and Clarius HD3 etc.) currently used in routine clinical practice.

SUMMARY:
Transcranial Ultrasound via Sonolucent Cranioplasty is a prospective, single arm, observational, open label (non-blinded) study to collect real world evidence on the use of transcranial ultrasound via sonolucent cranioplasty.

DETAILED DESCRIPTION:
Standard of care (SOC) imaging techniques routinely used for neurosurgical monitoring, namely computed tomography (CT) and magnetic resonance imaging (MRI), present numerous patient, provider, and institutional burdens associated with transport, invasiveness, contrast administration, radiation exposure, imaging delay, and overall global costs. Ultrasound represents a promising alternative that overcomes many of these disadvantages being noninvasive, low-risk, real-time and portable, but is limited by the acoustic impedance of autologous cranial bone. Recently, material innovations enabling both transparent and sonolucent polymethyl methacrylate (PMMA) - a material commonly used for cranial reconstruction with a longstanding history of safety - have facilitated ultrasound windows within patients already receiving cranioplasty as standard of care. Early results applying transcranioplasty ultrasound (TCUS) through sonolucent cranial plates have been encouraging in regard to agreement with SOC imaging and advanced doppler capabilities. That said, limited published data exists commensurate with the novelty of the technique, therefore investigators herein aim to address this paucity by investigating the feasibility and efficacy of TCUS as compared to standard of care postoperative imaging modalities (i.e. MRI & CT) in a prospective, quality control study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Patients who are undergoing reconstructive sonolucent cranioplasty as standard of care.
4. Male or female, aged ≥ 18.

Exclusion Criteria:

1. Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Neuroanatomy accuracy of TCUS | 12 months
  Accuracy metrics related to identification and measurement of neuroanatomy structures using Trasncranial Ultrasound
Diagnostic accuracy of TCUS | 12 months
  Accuracy metrics related to detection of postoperative complications using Trasncranial Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Netanel Ben-Shalom, MD, Principal Investigator — Lenox Hill Hospital
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No